CLINICAL TRIAL: NCT05742984
Title: A Phase 1, Open Label, Randomized, Parallel-group, Single Center Study to Investigate Pharmacokinetics and Pharmacodynamics (Intragastric pH) of Linaprazan Glurate/Linaprazan After Single and 14 Days'Repeated Oral Administration of Linaprazan Glurate to Healthy Subjects
Brief Title: Investigate Linaprazan Glurate/Linaprazan in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cinclus Pharma Holding AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX842A2107
Record Dates: First submitted 2023-01-02; First posted 2023-02-24 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: 25 mg linaprazan glurate QD (Experimental): 25 mg (one 25 mg oral tablet) linaprazan glurate once daily (QD) for 14 days
  Interventions: Drug: linaprazan glurate 25 mg QD
- Group 2: 50 mg Linaprazan Glurate QD (Experimental): 50 mg (two 25 mg oral tablets) linaprazan glurate once daily (QD) for 14 days
  Interventions: Drug: linaprazan glurate 50 mg QD
- Group 3: 75 mg Linaprazan Glurate QD (Experimental): 75 mg (three 25 mg oral tablet) linaprazan glurate once daily (QD) for 14 days
  Interventions: Drug: linaprazan glurate 75 mg QD
- Group 4: 25 mg Linaprazan Glurate BID (Experimental): 25 mg (one 25mg oral tablet) linaprazan glurate twice daily (BID) for 14 days
  Interventions: Drug: linaprazan glurate 25 mg BID
- Group 5: 50 mg Linaprazan Glurate BID (Experimental): 50 mg (two 25 mg oral tablets) linaprazan glurate twice daily (BID) for 14 days
  Interventions: Drug: linaprazan glurate 50 mg BID
- Group 6: 75 mg Linaprazan Glurate BID (Experimental): 75 mg (three 25 mg oral tablet) linaprazan glurate twice daily (BID) for 14 days
  Interventions: Drug: linaprazan glurate 75 mg BID

INTERVENTIONS:
Drug: linaprazan glurate 25 mg QD — The subjects will receive 25 mg dose in the evening, in a non-fasted condition 30 minutes after the evening meal, for 14 days. Subjects are to follow a standardized food intake schedule.
  After a drug holiday period of either 2, 4 or 6 days, linaprazan glurate will be given once more in the evening (non-fasted).
  Arms: Group 1: 25 mg linaprazan glurate QD
Drug: linaprazan glurate 50 mg QD — The subjects will receive 50 mg dose in the evening, in a non-fasted condition 30 minutes after the evening meal, for 14 days. Subjects are to follow a standardized food intake schedule.
  After a drug holiday period of either 2, 4 or 6 days, linaprazan glurate will be given once more in the evening (non-fasted).
  Arms: Group 2: 50 mg Linaprazan Glurate QD
Drug: linaprazan glurate 75 mg QD — The subjects will receive 75 mg dose in the evening, in a non-fasted condition 30 minutes after the evening meal, for 14 days. Subjects are to follow a standardized food intake schedule.
  After a drug holiday period of either 2, 4 or 6 days, linaprazan glurate will be given once more in the evening (non-fasted).
  Arms: Group 3: 75 mg Linaprazan Glurate QD
Drug: linaprazan glurate 25 mg BID — The subjects will receive 25 mg dose twice daily, in the morning and in the evening for 14 days. Subjects will be fasted for ≥10 hours overnight before dosing on Day 1 and day 14, until 30 minutes post-dose. During fasting, tap water, but no other drinks, are allowed as desired, except for 1 hour before and 30 minutes after dosing. The second daily dose will be administered 30 minutes after the evening meal, i.e. in a non-fasted condition. The subjects are to follow a standardized food intake schedule. After a drug holiday period of either 2, 4 or 6 days, linaprazan glurate will be given once more (in fasted condition in the morning, non-fasted in the evening).
  Arms: Group 4: 25 mg Linaprazan Glurate BID
Drug: linaprazan glurate 50 mg BID — The subjects will receive 50 mg dose twice daily, in the morning and in the evening for 14 days. Subjects will be fasted for ≥10 hours overnight before dosing on Day 1 and day 14, until 30 minutes post-dose. During fasting, tap water, but no other drinks, are allowed as desired, except for 1 hour before and 30 minutes after dosing. The second daily dose will be administered 30 minutes after the evening meal, i.e. in a non-fasted condition. The subjects are to follow a standardized food intake schedule. After a drug holiday period of either 2, 4 or 6 days, linaprazan glurate will be given once more (in fasted condition in the morning, non-fasted in the evening).
  Arms: Group 5: 50 mg Linaprazan Glurate BID
Drug: linaprazan glurate 75 mg BID — The subjects will receive 75 mg dose twice daily, in the morning and in the evening for 14 days. Subjects will be fasted for ≥10 hours overnight before dosing on Day 1 and day 14, until 30 minutes post-dose. During fasting, tap water, but no other drinks, are allowed as desired, except for 1 hour before and 30 minutes after dosing. The second daily dose will be administered 30 minutes after the evening meal, i.e. in a non-fasted condition. The subjects are to follow a standardized food intake schedule. After a drug holiday period of either 2, 4 or 6 days, linaprazan glurate will be given once more (in fasted condition in the morning, non-fasted in the evening).
  Arms: Group 6: 75 mg Linaprazan Glurate BID

SUMMARY:
This is a Phase I, single-center, open label parallel-group, randomized study designed to evaluate the pharmacokinetics (PK), pharmacodynamics (PD, by continuous intragastric pH measurment), safety and tolerability of single and repeated oral doses of linaprazan glurate in 3 different dose levels given once- (QD) or twice daily (BID), for 14 days, with an additional single dose after 2, 4 or 6 days of drug holiday. The population will include healthy male and female subjects.

The subjects will be followed up to 28 days post IMP dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female subject aged 18 to 65 years, inclusive.
3. Body mass index ≥ 18.5 and ≤ 30.0 kg/m2.
4. Medically healthy, without abnormal clinically significant medical history, physical findings, vital signs, ECGs, or laboratory values at the time of screening, as judged by the Investigator.

Exclusion Criteria:

1. Female subjects of childbearing potential (defined as all subjects physiologically capable of becoming pregnant)
2. Male subjects with a partner of childbearing potential
3. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
4. History of GERD or clinically significant acid reflux, as judged by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Turk, M.Pharm, Study Director — CRS d.o.o Ljubljana, Ukmarjeva Ulica 6, Slovenia, 1000 Contact: Tanja Turk, M.pharm +38651619388 tanja.turk@crs.si
Locations (1):
- CRS d.o.o,Ukmarjeva ulica 6, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 132 subjects were screened, of which 75 subjects were randomized, including 2 subjects who did not receive any study medication. Hence 73 subjects were randomized and received at least 1 dose of linaprazan glurate. Three subjects withdrew consent and 3 subjects discontinued due to adverse AEs. A total of 69 subjects completed the study.
Groups:
- 25 mg Linaprazan Glurate QD: 25 mg ( one 25 mg oral tablet) Linaprazan Glurate QD for 14 days
  Linaprazan Glurate 25 mg: The participating subjects will receive 25 mg doses of IMP, QD or BID for 14 days. After a drug holiday period (2, 4 or 6 days), linaprazan glurate will be given once more (QD or BID, on Day 16, 18 or 20). In total, 15 or 30 doses will be given.
- 50 mg Linaprazan Glurate QD: 50 mg (two 25 mg oral tablets) Linaprazan Glurate QD for 14 days
  Linaprazan Glurate 50 mg: The participating subjects will receive 50 mg doses of IMP, QD or BID for 14 days. After a drug holiday period (2, 4 or 6 days), linaprazan glurate will be given once more (QD or BID, on Day 16, 18 or 20). In total, 15 or 30 doses will be given.
- 75 mg Linaprazan Glurate QD: 75 mg ( three 25 mg oral tablet) Linaprazan Glurate QD for 14 days
  Linaprazan Glurate 75 mg: The participating subjects will receive 75 mg doses of IMP, QD or BID for 14 days. After a drug holiday period (2, 4 or 6 days), linaprazan glurate will be given once more (QD or BID, on Day 16, 18 or 20). In total, 15 or 30 doses will be given.
- 25 mg Linaprazan Glurate BID: 25 mg ( one 25mg oral tablet) Linaprazan Glurate BID for 14 days
  Linaprazan Glurate 25 mg: The participating subjects will receive 25 mg doses of IMP, QD or BID for 14 days. After a drug holiday period (2, 4 or 6 days), linaprazan glurate will be given once more (QD or BID, on Day 16, 18 or 20). In total, 15 or 30 doses will be given.
- 50 mg Linaprazan Glurate BID: 50 mg ( two 25 mg oral tablets) Linaprazan Glurate BID for 14 days
  Linaprazan Glurate 50 mg: The participating subjects will receive 50 mg doses of IMP, QD or BID for 14 days. After a drug holiday period (2, 4 or 6 days), linaprazan glurate will be given once more (QD or BID, on Day 16, 18 or 20). In total, 15 or 30 doses will be given.
- 75 mg Linaprazan Glurate BID: 75 mg ( three 25 mg oral tablet) Linaprazan Glurate BID for 14 days
  Linaprazan Glurate 75 mg: The participating subjects will receive 75 mg doses of IMP, QD or BID for 14 days. After a drug holiday period (2, 4 or 6 days), linaprazan glurate will be given once more (QD or BID, on Day 16, 18 or 20). In total, 15 or 30 doses will be given.
Period: Overall Study
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID
Started | 12 | 13 | 13 | 12 | 12 | 13
Completed | 12 | 12 | 12 | 12 | 11 | 10
Not Completed | 0 | 1 | 1 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 25 mg Linaprazan Glurate QD: 25 mg (one 25 mg oral tablet) linaprazan glurate QD for 14 days
- 50 mg Linaprazan Glurate QD: 50 mg (two 25 mg oral tablets) linaprazan glurate QD for 14 days
- 75 mg Linaprazan Glurate QD: 75 mg (three 25 mg oral tablets) linaprazan glurate QD for 14 days
- 25 mg Linaprazan Glurate BID: 25 mg (one 25mg oral tablet) linaprazan glurate BID for 14 days
- 50 mg Linaprazan Glurate BID: 50 mg (two 25 mg oral tablets) linaprazan glurate BID for 14 days
- 75 mg Linaprazan Glurate BID: 75 mg (three 25 mg oral tablets) linaprazan glurate BID for 14 days
- Total: Total of all reporting groups
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID | Total
Number analyzed (Participants) | 12 | 13 | 13 | 12 | 11 | 12 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (8.26) | 24.7 (8.35) | 22.8 (2.45) | 22.4 (1.88) | 23.9 (3.48) | 25.1 (8.25) | 23.8 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 5 | 5 | 5 | 32
  Male | 7 | 7 | 7 | 7 | 6 | 7 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 13 | 13 | 12 | 11 | 12 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 12 | 13 | 13 | 12 | 11 | 12 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Slovenia | 12 | 13 | 13 | 12 | 11 | 12 | 73

OUTCOME MEASURES:

1. Primary Outcome: AUC0-24h Linaprazan (QD)
Description: Linaprazan area under the plasma concentration curve, from 0 to 24h post dose on Day 1 and Day 14. QD groups only.
Time Frame: Day 1 and Day 14
Population: Overall # of participants analyzed does not match the participant flow figures due a discrepancy between "completers" and "evaluable" participants (protocol deviations). Figures here represent the number of evaluable subjects.
  NB! One participant in 50mg QD discontinued before completion of the full study, but only after the primary variables had been collected. Thus this participant's data was evaluable despite being a non-completer.
Measure: Mean (Standard Deviation); unit: nmol/L*h
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD
Number analyzed (Participants) | 12 | 13 | 12
nmol/L*h
  AUC0-24h Day 1 | 5057 (1650.6) | 8924 (2281.0) | 13900 (4339.5)
  AUC0-24h Day 14 | 4640 (1657.4) | 8626 (3571.9) | 11697 (4053.3)

2. Primary Outcome: AUC0-12, 12-24h Linaprazan (BID)
Description: Linaprazan area under the plasma concentration curve, from 0 to 12h and 12-24h post dose on Day 1 and Day 14. BID groups only.
Time Frame: Day 1 and Day 14
Measure: Mean (Standard Deviation); unit: nmol/L*h
Arm/Group | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID
Number analyzed (Participants) | 12 | 11 | 10
nmol/L*h
  AUC0-12h Day 1 | 4081 (1351.9) | 8084 (1400.5) | 11814 (3181.8)
  AUC12-24h Day 1 | 3947 (939.8) | 7107 (1917.8) | 9532 (2118.1)
  AUC0-12h Day 14 | 4896 (1367.3) | 7518 (1627.0) | 11757 (3058.3)
  AUC12-24h Day 14 | 4002 (1142.8) | 6334 (2061.6) | 9609 (2087.5)

3. Primary Outcome: Cmax Linaprazan (QD)
Description: Linaprazan maximum plasma concentration 0-24h post dose for QD groups, at day 1 and day 14.
Time Frame: Day 1 and day 14
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD
Number analyzed (Participants) | 12 | 13 | 12
nmol/L
  Cmax day 1 | 527.5 (184.929) | 1066.23 (209.973) | 1594.42 (585.525)
  Cmax day 14 | 404.75 (174.068) | 1002.00 (538.574) | 1044.92 (478.102)

4. Primary Outcome: Cmax Linaprazan (BID)
Description: Linaprazan maximum plasma concentration 0-12h, and 12-24h post dose for BID groups, at day 1 and day 14.
Time Frame: Day 1 and day 14
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- 25 mg Linaprazan Glurate BID: 25 mg (one 25 mg oral tablet) linaprazan glurate BID for 14 days
Arm/Group | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID
Number analyzed (Participants) | 12 | 11 | 10
nmol/L
  Cmax 0-12h day 1 | 658.42 (212.101) | 1380.18 (303.283) | 1942.00 (667.280)
  Cmax 12-24h day 1 | 520.92 (126.378) | 997.09 (363.660) | 1283.90 (435.399)
  Cmax 0-12h day 14 | 782.92 (263.988) | 1148.64 (415.251) | 1740.60 (468.197)
  Cmax 12-24h day 14 | 520.83 (144.568) | 842.36 (270.396) | 1285.50 (443.703)

5. Primary Outcome: AUC0-24h Linaprazan Glurate (QD)
Description: Linaprazan glurate area under the plasma concentration curve, from 0-24h post dose on Day 1 and Day 14. QD groups only.
Time Frame: Day 1 and day 14
Measure: Mean (Standard Deviation); unit: nmol/L*h
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD
Number analyzed (Participants) | 12 | 13 | 12
nmol/L*h
  AUC0-24h Day 1 | 42 (18.9) | 99 (68.0) | 166 (85.5)
  AUC0-24h Day 14 | 27 (18.6) | 107 (97.9) | 149 (201.1)

6. Primary Outcome: AUC0-12h, 12-24h Linaprazan Glurate (BID)
Description: Linaprazan glurate area under the plasma concentration curve, from 0 to 12h and 12-24h post dose on Day 1 and Day 14. BID groups only.
Time Frame: Day 1 and Day 14
Measure: Mean (Standard Deviation); unit: nmol/L*h
Arm/Group | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID
Number analyzed (Participants) | 12 | 11 | 10
nmol/L*h
  AUC0-12h Day 1 | 40 (15.5) | 117 (65.3) | 179 (87.4)
  AUC 12-24h Day 1 | 30 (14.6) | 74 (40.7) | 78 (24.7)
  AUC0-12h Day 14 | 39 (23.2) | 69 (37.0) | 156 (140.6)
  AUC 12-24h Day 14 | 28 (10.2) | 68 (38.1) | 114 (91.2)

7. Primary Outcome: Cmax Linaprazan Glurate (QD)
Description: Linaprazan glurate maximum plasma concentration 0-24h post dose for QD groups, at day 1 and day 14.
Time Frame: Day 1 and day 14
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- 25 mg Linaprazan Glurate QD: 25 mg (one 25mg oral tablet) linaprazan glurate QD for 14 days
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD
Number analyzed (Participants) | 12 | 13 | 12
nmol/L
  Cmax Day 1 | 27.54 (21.284) | 62.24 (53.653) | 100.46 (64.576)
  Cmax Day 14 | 18.43 (18.775) | 126.31 (166.828) | 107.07 (202.899)

8. Primary Outcome: Cmax Linaprazan Glurate (BID)
Description: Linaprazan glurate maximum plasma concentration 0-12h and 12-24h post dose for BID groups, at day 1 and day 14.
Time Frame: Day 1 and day 14
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID
Number analyzed (Participants) | 12 | 11 | 10
nmol/L
  Cmax0-12h Day 1 | 32.52 (19.704) | 101.26 (49.177) | 148.19 (80.799)
  Cmax 12-24h Day 1 | 14.69 (10.290) | 46.60 (40.041) | 40.41 (32.422)
  Cmax0-12h Day 14 | 47.59 (46.275) | 61.09 (43.234) | 151.73 (145.527)
  Cmax 12-24h Day 14 | 22.29 (13.414) | 41.51 (38.110) | 94.42 (140.218)

9. Primary Outcome: Percentage of Time Gastric pH >4 Over a 24-hour Monitoring Period (Holding Time Ratio, HTR)
Description: Percentage of time gastric pH >4 at Days 1 and 14 over a 24-hour monitoring period following linaprazan glurate administration.
  Intragastric pH was measured every second with an intragastric probe. The measurements were compressed into 10-minute median intervalls before calculating the % of time with intragastric >pH 4 (HTR). The HTR is presented with descriptive statistics, by dosing group.
Time Frame: Day 1 and day 14
Population: PK/PD analysis set (PK/PDAS), a subset of the PK-analysis set, included all pH measurements which were evaluable. 4 subjects were excluded from the PK-analysis set, and thereby also from the PK/PDAS subset, due to study drug incompliance. Another 5 subjects were excluded entirely from the PK/PDAS due to presence of H. pylori (exclusion criteria - could have an impact on acid suppression sensitivity). In total 67 individuals provided at least 1 evaluable pH curve.
Measure: Mean (Standard Deviation); unit: % of time
Groups:
- 25 mg Linaprazan Glurate QD: The subjects received 25 mg dose in the evening, in a non-fasted condition 30 minutes after the evening meal, for 14 days. Subjects followed a standardized food intake schedule.
- 50 mg Linaprazan Glurate QD: The subjects received 50 mg dose in the evening, in a non-fasted condition 30 minutes after the evening meal, for 14 days. Subjects followed a standardized food intake schedule.
- 75 mg Linaprazan Glurate QD: The subjects received 75 mg dose in the evening, in a non-fasted condition 30 minutes after the evening meal, for 14 days. Subjects followed a standardized food intake schedule.
- 25 mg Linaprazan Glurate BID: The subjects will received 25 mg dose twice daily, in the morning and in the evening for 14 days. Subjects were fasted for ≥10 hours overnight before dosing on Day 1 and day 14, until 30 minutes post-dose. During fasting, tap water, but no other drinks, were allowed as desired, except for 1 hour before and 30 minutes after dosing.
  The second daily dose was administered 30 minutes after the evening meal, i.e. in a non-fasted condition. The subjects followed a standardized food intake schedule.
- 50 mg Linaprazan Glurate BID: The subjects will received 50 mg dose twice daily, in the morning and in the evening for 14 days. Subjects were fasted for ≥10 hours overnight before dosing on Day 1 and day 14, until 30 minutes post-dose. During fasting, tap water, but no other drinks, were allowed as desired, except for 1 hour before and 30 minutes after dosing.
  The second daily dose was administered 30 minutes after the evening meal, i.e. in a non-fasted condition. The subjects followed a standardized food intake schedule.
- 75 mg Linaprazan Glurate BID: The subjects will received 75 mg dose twice daily, in the morning and in the evening for 14 days. Subjects were fasted for ≥10 hours overnight before dosing on Day 1 and day 14, until 30 minutes post-dose. During fasting, tap water, but no other drinks, were allowed as desired, except for 1 hour before and 30 minutes after dosing.
  The second daily dose was administered 30 minutes after the evening meal, i.e. in a non-fasted condition. The subjects followed a standardized food intake schedule.
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID
Number analyzed (Participants) | 12 | 12 | 13 | 9 | 11 | 10
% of time
  HTR (%) pH >4 day 1 | 48 (23.23) | 64.6 (13.33) | 68.1 (23.48) | 76.0 (13.52) | 87.4 (8.62) | 94.5 (4.18)
  HTR (%) pH >4 day 14: number analyzed (Participants) | 12 | 12 | 11 | 9 | 11 | 8
  HTR (%) pH >4 day 14 | 48.5 (30.62) | 63.9 (20.09) | 87.2 (11.44) | 76.9 (20.13) | 95.7 (5.55) | 99.0 (1.54)

ADVERSE EVENTS:
Time Frame: (S)AE collection was performed on all dosed subjects, in the timeframe between first dose and until safety follow-up 7 +/-2 days after last dose, totalling ca 23-30 days of safety data collection. There was an exception made in the collection timeframe for the SAE, which occurred approximately 2 hours prior to first dose, i.e. outside the actual AE collection time frame as defined by the protocol, but since the event was deemed study procedure related it was reported as an SAE nevertheless.
Description: AEs were coded using MedDRA® Version 25.0. Verbatim terms were coded to lower-level terms within the primary SOC. All AEs reported are MedDRA PTs unless stated otherwise. During the study, the iSRC had 4 meetings to oversee the safety of each subject and all aggregate safety data was reviewed at each meeting.
  Number of participants in the All cause mortality and SAE fields below relate to all dosed participants (safety analysis set).
Groups:
- 50 mg Linaprazan Glurate BID: 50 mg ( two 25 mg oral tablets) linaprazan glurate BID for 14 days
Arm/Group | 25 mg Linaprazan Glurate QD | 50 mg Linaprazan Glurate QD | 75 mg Linaprazan Glurate QD | 25 mg Linaprazan Glurate BID | 50 mg Linaprazan Glurate BID | 75 mg Linaprazan Glurate BID
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/12 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/13 | 0/12 | 0/11 | 1/12
Other Adverse Events (participants affected / at risk) | 6/12 | 8/13 | 6/13 | 7/12 | 6/11 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg Linaprazan Glurate QD (N=12) | 50 mg Linaprazan Glurate QD (N=13) | 75 mg Linaprazan Glurate QD (N=13) | 25 mg Linaprazan Glurate BID (N=12) | 50 mg Linaprazan Glurate BID (N=11) | 75 mg Linaprazan Glurate BID (N=12)
Commotio cerebri (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — not related to the IMP and probably related to the study procedure of blood sampling.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg Linaprazan Glurate QD (N=12) | 50 mg Linaprazan Glurate QD (N=13) | 75 mg Linaprazan Glurate QD (N=13) | 25 mg Linaprazan Glurate BID (N=12) | 50 mg Linaprazan Glurate BID (N=11) | 75 mg Linaprazan Glurate BID (N=12)
Headache (Nervous system disorders) | 3 (6) | 3 (5) | 1 (1) | 3 (3) | 3 (3) | 3 (5)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post streptoccocal glumerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial Bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
arterial puncture (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT05742984/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT05742984/SAP_001.pdf